CLINICAL TRIAL: NCT00533832
Title: A Multicernter, Pivotal, Safety and Efficacy Study of the NeuroCtybernetic Prosthesis (NCP(R)) System in Patients With Depression
Brief Title: Pivotal Trial (D02) of Vagus Nerve Stimulation (VNS) for Treatment-Resistant Depression (TRD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyberonics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D02
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Last update posted 2007-09-24 (Estimated); Status verified 2007-09

CONDITIONS: Major Depressive Disorder
Keywords: depression; vagus nerve stimulation
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Patients implanted with the vagus nerve stimulation (VNS) device and receiving VNS Intervention: vagus nerve stimulation (VNS)
  Interventions: Device: vagus nerve stimulation (VNS)
- 2 (Placebo Comparator): Implanted with vagus nerve stimulation (VNS) device, but not receiving VNS
  Interventions: Device: vagus nerve stimulation (VNS)

INTERVENTIONS:
Device: vagus nerve stimulation (VNS) — intermittent vagus nerve stimulation
  Placebo group were implanted, but did not receive vagus nerve stimulation during the acute phase.

SUMMARY:
To confirm the safety and efficacy of the NCP System in treating patients in a nmajor depressive episode.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with major depressive episode (MDE)
2. chronic (>=2 years)or recurrent (>-=4) lifetime MDEs
3. resistant to >=2 treatments from different categories
4. completed >=6 weeks of psychotherapy
5. score >=20 on 24-item Hamilton Rating Scale of Depression
6. IQ >=70
7. stable on current antidepressant medication (no more than 5 antidepressant meds) or taking no antidepressant meds for >=4 weeks before Visit B1
8. stable on atypical antipsychotic and anticonvulsant medications as for item #7
9. age >=18 amd <=80 years
10. male or nonpregnant female adequately protected from conception.
11. able to comply with testing and follow-up visits
12. voluntarily signed informed consent
13. patients with bipolar disorder demonstrated a resistance to lithium treatment or has a medical contraindication to treatment with lithium or is known to be intolerant to lithium (not applicable to patients with MDD)

Exclusion Criteria:

1. atypical depression at study entry or psychotic symptoms in any MDE
2. history of schizophrenia, schizoaffective disorder, or delusional disorders
3. rapid cycling bopolar disorder
4. secondary diagnosis of, or signs of, delirium, dementia, amnestic, or other cognitive disorders
5. failed 7 or more antidepressant treatments
6. a. suicide attempt requiring medical attention within previous 12 months b. >=2 suicide attempts in the past 12 months c. cannot guarantee that will not implement suicide d. likely to attempt suicide within next 6 mon in investigator's opinion
7. alcohol or substance dependence within previous 12 months or abuse within previous 6 mon other than nicotine dependence or abuse
8. history of myocardial infarction or cardiac arrest
9. other progressive neurological disease, significant central nervous system disease or injury, or cervical fracture that makes implantation difficult
10. received general anesthesia with 390 days before enrollment.
11. taken an investigational drug within a clearance duration of 5 x the half-life of the investigational drug or within <=4weeks before Visit B1, whichever time is greater
12. enrolled in another investigational study
13. using another investigational device
14. significant cardiac or pulmonary condition currently under treatment resulting in an ASA score >=III
15. history of, or evidence of, significant brain malformation or significant head injury or clinically apparent cerebral vascular events, or prior brain surgery such as cingulatomy
16. unilateral or bilateral cervical vagotomy
17. demand cardiac pacemaker, implantable defibrillator, or other implantable stimulator
18. likely to require a whole body MRI after NCP implantation
19. currently receiving or likely to receive short-wave diathermy, microwave diathermy, or therapeutic ultrasound diathermy after implantation
20. plans to relocate or move to a location distant from the study site within one year of enrollment
21. previously enrolled in this or any other NCP System study -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2000-07; Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Investigator, Study Director — Cyberonics, Inc.
Locations (1):
- Houston, Texas, United States

REFERENCES:
- [Result] George MS, Rush AJ, Marangell LB, Sackeim HA, Brannan SK, Davis SM, Howland R, Kling MA, Moreno F, Rittberg B, Dunner D, Schwartz T, Carpenter L, Burke M, Ninan P, Goodnick P. A one-year comparison of vagus nerve stimulation with treatment as usual for treatment-resistant depression. Biol Psychiatry. 2005 Sep 1;58(5):364-73. doi: 10.1016/j.biopsych.2005.07.028. PMID 16139582
- [Result] Rush AJ, Sackeim HA, Marangell LB, George MS, Brannan SK, Davis SM, Lavori P, Howland R, Kling MA, Rittberg B, Carpenter L, Ninan P, Moreno F, Schwartz T, Conway C, Burke M, Barry JJ. Effects of 12 months of vagus nerve stimulation in treatment-resistant depression: a naturalistic study. Biol Psychiatry. 2005 Sep 1;58(5):355-63. doi: 10.1016/j.biopsych.2005.05.024. PMID 16139581
- [Result] Rush AJ, Marangell LB, Sackeim HA, George MS, Brannan SK, Davis SM, Howland R, Kling MA, Rittberg BR, Burke WJ, Rapaport MH, Zajecka J, Nierenberg AA, Husain MM, Ginsberg D, Cooke RG. Vagus nerve stimulation for treatment-resistant depression: a randomized, controlled acute phase trial. Biol Psychiatry. 2005 Sep 1;58(5):347-54. doi: 10.1016/j.biopsych.2005.05.025. PMID 16139580
- [Derived] Cohen LJ, Allen JC Jr. Estimating the potential savings with vagus nerve stimulation for treatment-resistant depression: a payer perspective. Curr Med Res Opin. 2008 Aug;24(8):2203-17. doi: 10.1185/03007990802229050. PMID 18786301
- [Derived] Nierenberg AA, Alpert JE, Gardner-Schuster EE, Seay S, Mischoulon D. Vagus nerve stimulation: 2-year outcomes for bipolar versus unipolar treatment-resistant depression. Biol Psychiatry. 2008 Sep 15;64(6):455-60. doi: 10.1016/j.biopsych.2008.04.036. Epub 2008 Jun 24. PMID 18571625